CLINICAL TRIAL: NCT05268107
Title: Ethnic Differences in Mechanisms of Action of Dupilumab
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Johann E Gudjonsson MD PhD, Professor of Dermatology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00201405/Derm 759
Record Dates: First submitted 2022-02-22; First posted 2022-03-07 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis
Keywords: Asian patients; African American patients; Caucasian patients; Inflammatory responses; Dupixent; Dupilumab
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: A total of 10 Caucasian, 10 Asian (Eastern and Southeastern Asian), and 10 African American patients with moderate-to severe AD (5 males and 5 females in each group) will be enrolled.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dupilumab (Experimental): The 3 groups of patients (Asian, African American, and Caucasian) will all receive the same intervention.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Patients will be treated with dupilumab for 4 months (standard FDA-approved dosing of 600 mg subcutaneously at baseline/week 0, followed by 300 mg every 2 weeks).
  Skin biopsies will be assessed at baseline (lesional and non-lesional), week 2 (lesional), and week 16 (lesional). In addition, blood will be obtained at baseline and week 16.
  Other Names: Dupixent

SUMMARY:
Previous research has shown that Asian and African Americans are more likely to develop atopic dermatitis (AD) than their Caucasian counterparts. However, limited information is known about AD in Asian and African American populations because most molecular studies have focused on Caucasians with AD.

This trial will determine differences in inflammatory responses to dupilumab between Caucasian, Asian, and African American patients with AD.

The central hypothesis of this study is that ethnic differences in both immune and stromal cells contribute to variability in AD presentation and response to anti-interleukin-4 receptor (IL-4R) inhibition with dupilumab.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of AD for at least 2 years before the screening visit and confirmed according to the American Academy of Dermatology Consensus Criteria at the time of the screening visit
* Moderate-to-severe AD with involvement > 10% of body-surface-area (BSA) and investigator global assessment (IGA) score 3 (based on the IGA scale ranging from 0 to 4, in which 3 is moderate and 4 is severe) at both the screening and baseline visits
* Female subjects of childbearing potential (i.e., fertile, following menarche and until becoming post-menopausal unless permanently sterile) must agree either to commit to true abstinence throughout the study and for 12 weeks after the last study drug injection or to use an adequate and approved method of contraception throughout the study and for 12 weeks after the last study drug injection
* Subject willing and able to comply with all of the time commitments and procedural requirements of the clinical study protocol

Exclusion Criteria:

* Body weight less than 30 kilogram
* Subjects meeting 1 or more of the following criteria at screening or baseline:

  1. Had an exacerbation of asthma requiring hospitalization in the preceding 12 months.
  2. Reporting asthma that has not been well-controlled (ie, symptoms occurring on >2 days per week, nighttime awakenings 2 or more times per week, or some interference with normal activities) during the preceding 3 months
  3. Asthma Control Test (ACT) < 19 (only for subjects with a history of asthma).
  4. Subjects with a current medical history of chronic obstructive pulmonary disease and/or chronic bronchitis.
* Cutaneous infection within 1 week before the baseline visit, any infection requiring treatment with oral or parenteral antibiotics, antivirals, antiparasitics, or antifungals within 2 weeks before the baseline visit.
* Confirmed or suspected coronavirus disease 2019 (COVID-19) infection within 4 weeks before the screening or baseline visit
* Received COVID-19 vaccination within 4 weeks before baseline visit
* Previous treatment with dupilumab
* Pregnant women (positive serum pregnancy test result at the screening visit or positive urine pregnancy test at the baseline visit), breastfeeding women, or women planning a pregnancy during the clinical study
* History of lymphoproliferative disease or history of malignancy of any organ system within the last 5 years, except for basal cell carcinoma, squamous cell carcinoma in situ (Bowen's disease), or carcinomas in situ of the cervix that have been treated and have no evidence of recurrence in the last 12 weeks before the baseline visit
* History of hypersensitivity (including anaphylaxis) to an immunoglobulin product (plasma-derived or recombinant, i.e., monoclonal antibody) or to lidocaine
* Known active or latent tuberculosis (TB) infection
* Known or suspected immunosuppression or unusually frequent, recurrent, severe, or prolonged infections as per investigator judgment
* History of or current confounding skin condition (i.e., Netherton syndrome, psoriasis, cutaneous T-cell lymphoma [mycosis fungoides or Sezary syndrome], contact dermatitis, chronic actinic dermatitis, dermatitis herpetiformis)
* Planned or expected major surgical procedure during the study
* Currently participating or participated in any other study of a drug or device, within the past 8 weeks before the screening visit, or is in an exclusion period (if verifiable) from a previous study
* History of alcohol or substance abuse within 6 months of the screening
* History of poor wound healing or keloid formation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Difference in inflammatory response to dupilumab between Caucasian, Asian and African American patients with atopic dermatitis as measured by change in expression of interleukin4 (IL4) from week 0 to 2. | Week 0, week 2

SECONDARY OUTCOMES:
Difference in inflammatory response to dupilumab between Caucasian, Asian and African American patients with atopic dermatitis as measured by change in expression of interleukin13 from week 0 to 2. | Week 0, week 2
Difference in inflammatory response to dupilumab between Caucasian, Asian and African American patients with atopic dermatitis as measured by change in expression of Interferon (IFN) from week 0 to 2. | Week 0, week 2
Difference in inflammatory response to dupilumab between Caucasian, Asian and African American patients with atopic dermatitis as measured by change in expression of interleukin36 from week 0 to 2. | Week 0, week 2
Difference in inflammatory response to dupilumab between Caucasian, Asian and African American patients with atopic dermatitis as measured by change in expression of interleukin4 from week 0 to 16. | Week 0 to week 16
Difference in inflammatory response to dupilumab between Caucasian, Asian and African American patients with atopic dermatitis as measured by change in expression of interleukin13 from week 0 to 16. | Week 0 to week 16
Difference in inflammatory response to dupilumab between Caucasian, Asian and African American patients with atopic dermatitis as measured by change in expression of IFN from week 0 to 16. | Week 0 to week 16
Difference in inflammatory response to dupilumab between Caucasian, Asian and African American patients with atopic dermatitis as measured by change in expression of interleukin36 from week 0 to 16. | Week 0 to week 16

CONTACTS AND LOCATIONS:
Overall Officials: Johann Gudjonsson, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No